CLINICAL TRIAL: NCT03284359
Title: A Randomized Trial of Nudges To Enhance Enrollment in Critical Care Research
Brief Title: Use of Nudges To Enhance Enrollment in Critical Care Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 828046
Record Dates: First submitted 2017-08-15; First posted 2017-09-15 (Actual); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Critical Illness
Keywords: Critical Illness; Mechanical Ventilation; Economics, Behavioral; Surrogate decision maker
MeSH Terms: conditions — Critical Illness; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Consent Nudge Bundle (Experimental): Arm 1 will be administered a novel pre-consent nudge bundle which incorporates several behavioral economic interventions within a brief survey. Participants will subsequently be asked by the same research personnel to participate in a simulated randomized control trial (RCT) comparing two mechanical ventilation weaning protocols among mechanically ventilated patients. Participants will receive the standard consent form followed by a risk assessment and demographic survey.
  Interventions: Behavioral: Pre-Consent Nudge Bundle
- Standard Consent (No Intervention): Arm 2 will serve as the control arm. Participants will be approached by the research personnel to participate in a simulated RCT comparing two mechanical ventilation weaning protocols among mechanically ventilated patients. Participants will receive a standard consent form as detailed in the Study Instruments section. Following the consent process participants will conduct the same risk assessment survey and demographic survey.

INTERVENTIONS:
Behavioral: Pre-Consent Nudge Bundle — The pre-consent nudge bundle survey was developed by the study team and incorporates several behavioral interventions into a bundle of 5 types of nudges: (i) injunctive norms; (ii) descriptive norms; (iii) duty of reciprocity; (iv) self-prophecy; and (v) foot-in-the-door. Injunctive norms involve the perception of what behavior is acceptable, while descriptive norms highlight what behaviors others are engaging in. The duty of reciprocity is the sense that one should repeat pro-social behavior for which they have benefited from. The foot-in-the-door nudge involves asking a participant to perform a small request which has a high consent rate followed by a larger request. The bundle consists of six questions and one statement.
  Arms: Pre-Consent Nudge Bundle

SUMMARY:
Difficulties enrolling patients in randomized clinical trials (RCTs) have long been recognized as a major barrier to successful evaluation of medical interventions. This is particularly problematic among intensive care unit (ICU) trials, of which more than one-third do not reach target enrollment. Under-enrollment and selective enrollment reduce RCTs' abilities to answer the research questions, thereby degrading the trials' scientific value and ethics.

Current evidence suggests that financial incentives can ethically increase study enrollment, but this approach can pose large up-front costs to researchers. However, several nonmonetary behavioral interventions, or nudges, may offer novel and easily scalable approaches to increase enrollment in RCTs.

The investigation team propose a 2-arm RCT in 10 ICUs at Penn to test the relative effectiveness of nudges on enrollment rates. Investigators hypothesize that a bundle of nudges during recruitment will increase enrollment rates compared to usual recruitment procedures will increase enrollment.

Investigators will enroll 182 critically ill patients' surrogate decision makers(participants) to engage in recruitment procedures for a simulated RCT comparing two mechanical ventilation weaning protocols among mechanically ventilated patients. Investigators will also measure participants' assessment of risk of the simulated trial after the informed consent process. This work will provide the first empirical evidence regarding the efficacy of inexpensive, scalable nudges to potentially augment enrollment and reduce costs of future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Surrogate decision-makers of patients who are:

1. Patient and surrogate is 18 years of age or older
2. Surrogate is English-proficient
3. Patient is mechanically ventilated
4. Patient is admitted to participating ICU

Exclusion Criteria:

Surrogate decision-makers of patients who are:

1. Patient is receiving comfort care only
2. Patient has anticipated extubation in the next 24 hours.
3. Patient with tracheostomy.
4. Bedside clinician declines patient participation.
5. Surrogate decision maker not available to approach prior to patient being extubated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Courtright, M.D., M.S., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krutsinger DC, O'Leary KL, Ellenberg SS, Cotner CE, Halpern SD, Courtright KR. A Randomized Controlled Trial of Behavioral Nudges to Improve Enrollment in Critical Care Trials. Ann Am Thorac Soc. 2020 Sep;17(9):1117-1125. doi: 10.1513/AnnalsATS.202003-194OC. PMID 32441987

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-Consent Nudge Bundle | Standard Consent
Started | 93 | 89
Completed | 93 | 89
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention to treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-Consent Nudge Bundle | Standard Consent | Total
Number analyzed (Participants) | 93 | 89 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (13.6) | 58.6 (17.2) | 60 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 58 | 53 | 111
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 23 | 38
  White | 74 | 59 | 133
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 7 | 11
Length of ICU stay at enrollment [Mean (Standard Deviation); unit: Hours] | 97.8 (73.1) | 114.5 (90.6) | 106.2 (81.9)

OUTCOME MEASURES:

1. Primary Outcome: Consent Rate
Description: The primary outcome is consent rate for a simulated RCT. This is an easily measurable binary outcome that has the potential for significant impact on future trial recruitment.
Time Frame: Up to 96 hours
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Consent Nudge Bundle | Standard Consent
Number analyzed (Participants) | 93 | 89
Participants | 27 | 30

2. Secondary Outcome: Risk Assessment
Description: Secondarily we will quantitatively assess the participant's assessment of the risk of participating in the simulated RCT. The risk assessment tool has been previously used in the assessment of risk perception of RCT participation in the setting of behavioral economic nudges. The risk assessment will be used to evaluate participants' impressions of the risk of participating in the RCT using a Likert scale ranging from 1 (Not risky at all) to 7 (very risky), as well as 9 comparative questions, each of which asks whether a study procedure was riskier than another risky activity, such as talking on one's cell phone while driving.
Time Frame: Up to 96 hours
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pre-Consent Nudge Bundle | Standard Consent
Number analyzed (Participants) | 93 | 89
units on a scale | 2 [0 to 5] | 2 [0 to 5.5]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the interaction. Long term adverse events were not evaluated.
Arm/Group | Pre-Consent Nudge Bundle | Standard Consent
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/89
Other Adverse Events (participants affected / at risk) | 0/93 | 0/89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03284359/Prot_SAP_ICF_000.pdf